CLINICAL TRIAL: NCT05328921
Title: Effects of Two Systemic Drugs on Intraocular Pressure in Narrow Angle Glaucoma
Brief Title: Effects of Systemic Drugs on Intraocular Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: Rc 9-22
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma, Angle-Closure; Glaucoma Suspect; Glaucoma Secondary to Drugs, Bilateral; Hypertension
Keywords: Angle closure glaucoma; Hypertension; Antihistaminic; Antihypertensive
MeSH Terms: conditions — Glaucoma, Angle-Closure; Ocular Hypertension; Hypertension | interventions — Antihypertensive Agents; Histamine Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Antihypertensive drugs group: Changes in IOP among patients on antihypertensive drugs
  Interventions: Drug: Antihypertensive Agents
- Antihistaminic drugs group: Changes in IOP among patients on antihistaminic drugs
  Interventions: Drug: Antihistaminics
- Antihypertensive and antihistaminic drugs group: Changes in IOP among patients on both antihypertensive and antihistaminic drugs
  Interventions: Drug: Antihypertensive Agents; Drug: Antihistaminics

INTERVENTIONS:
Drug: Antihypertensive Agents — Patients with narrow angle glaucoma and on systemic antihypertensive drugs.
  Groups: Antihypertensive and antihistaminic drugs group; Antihypertensive drugs group
Drug: Antihistaminics — Patients with narrow angle glaucoma and on systemic antihistaminic drugs.
  Groups: Antihistaminic drugs group; Antihypertensive and antihistaminic drugs group

SUMMARY:
To assess intraocular pressure changes among glaucoma patients on systemic antihypertensive and antihistaminic drugs.

DETAILED DESCRIPTION:
Changes in intraocular pressure in glaucomatous patients with narrow angle may elicit attacks of angle closure glaucoma.

In this study we aim to assess changes in intraocular pressure (IOP) among glaucomatous patients on systemic antihypertensive and antihistaminic drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients with narrow angle glaucoma on systemic antihypertensive and/or antihistaminic drugs.

Exclusion Criteria:

* open angle glaucoma patients confirmed by gonioscopy examination.
* Cases with dense corneal opacity or iris trauma that may affects gonioscopy examination.
* cases with secondary glaucoma.

Ages: 35 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients regularly visit glaucoma clinic at Banha university, EGYPT
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in intraocular pressure (IOP) measured by applanation tonometry | Immediately after visual acuity assessment for each eye after topical anesthetic eye drops and again on one and three months visit
  Changes in IOP measured by millimeter mercury (mmHg)

SECONDARY OUTCOMES:
Changes in pupil diameter | Immediately after slit lamp examination and again on one and three months visit
  Size of pupil measured in millimeters (mm) 7sing autorefractometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: Undecided